CLINICAL TRIAL: NCT05197387
Title: Inflammation in Intrahepatic Cholestasis of Pregnancy
Brief Title: Association of Intrahepatic Cholestasis of Pregnancy and Chronic Placental Inflammation
Acronym: INTREPIDE
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: INTREPIDE (29BRC21.0188)
Record Dates: First submitted 2022-01-05; First posted 2022-01-19 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Cholestasis of Pregnancy
Keywords: placenta; cholestasis; pregnancy; inflammation
MeSH Terms: conditions — Intrahepatic Cholestasis of Pregnancy; Cholestasis; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cases: Women with intrahepatic cholestasis of pregnancy
- Controls: Women without intrahepatic cholestasis of pregnancy

SUMMARY:
This observational prospective study will help to determine if an immune process similar to allograft rejection is responsible for the occurrence of an intrahepatic cholestasis of pregnancy (ICP).

If so, it would suggest the potential benefit of immunomodulatory therapeutics.

DETAILED DESCRIPTION:
This observational study will include 322 pregnant women at delivery: 161 women diagnosed with an intrahepatic cholestasis of pregnancy, and 161 control women.

A blood test will be performed at delivery for each woman and each newborn, in order to measure several biological parameters involved in inflammation processes, allograft rejection and angiogenesis. Placenta will also be analysed. In particular, we will look for chronic inflammation in placenta.

Biological parameters and placental parameters will be compared between the two groups: cases with ICP and controls.

ELIGIBILITY:
Inclusion Criteria:

* Adult pregnant woman with singleton

For cases: diagnosis of intrahepatic cholestasis of pregnancy For controls: no diagnosis of ICP

Exclusion Criteria:

* Women under 18 years old
* Women under legal protection
* Gemellar pregnancies
* Delivery before 22 Weeks of gestation
* Medical termination of pregnancy
* Acute chorioamniotitis, in particular those due to the following pathogens: toxoplasmosis, rubella, CMV, herpes virus
* Premature rupture of membranes <37SA
* Women infected by covid-19 in the month before delivery

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant woman
Study Population: Pregnant women with or without intrahepatic cholestasis of pregnancy included at delivery.
  Each control will be matched with each case according to gestation age at delivery.
Sampling Method: Probability Sample
Enrollment: 322 (Estimated)
Dates: Start 2022-06-21 (Actual); Primary Completion 2025-06-21 (Estimated); Study Completion 2025-06-22 (Estimated)

PRIMARY OUTCOMES:
Prevalence of placental chronic inflammation | At delivery

SECONDARY OUTCOMES:
Levels of several biological parameters involved in inflammation processes | At delivery
Levels of several biological parameters involved in allograft rejection | At delivery
Levels of several biological parameters involved in angiogenesis | At delivery

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - CHU Angers, Angers
  - Polyclinique KERAUDREN, Brest
  - CHU de Brest, Brest
  - CHU de Caen, Caen
  - CH de Chambery, Chambéry
  - CH Bretagne Sud, Lorient
  - CHU Nantes, Nantes
  - CH de Quimper, Quimper
  - CHU de Rennes, Rennes
  - CH St Brieuc, Saint-Brieuc
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning two years and ending five years following the publication
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.

REFERENCES:
- [Background] Du Q, Pan Y, Zhang Y, Zhang H, Zheng Y, Lu L, Wang J, Duan T, Chen J. Placental gene-expression profiles of intrahepatic cholestasis of pregnancy reveal involvement of multiple molecular pathways in blood vessel formation and inflammation. BMC Med Genomics. 2014 Jul 7;7:42. doi: 10.1186/1755-8794-7-42. PMID 25001852
- [Background] Patel S, Pinheiro M, Felix JC, Opper N, Ouzounian JG, Lee RH. A case-control review of placentas from patients with intrahepatic cholestasis of pregnancy. Fetal Pediatr Pathol. 2014 Aug;33(4):210-5. doi: 10.3109/15513815.2014.899413. Epub 2014 Apr 23. PMID 24758367
- [Background] Larson SP, Kovilam O, Agrawal DK. Immunological basis in the pathogenesis of intrahepatic cholestasis of pregnancy. Expert Rev Clin Immunol. 2016;12(1):39-48. doi: 10.1586/1744666X.2016.1101344. Epub 2015 Oct 15. PMID 26469633